CLINICAL TRIAL: NCT00224042
Title: A Randomized, Controlled, Open-label Study of the Safety and Efficacy of Ferrlecit® vs Oral Iron in Iron Deficient Patients With Chronic Kidney Disease Being Treated With Erythropoietic Therapy
Brief Title: Effect of Ferrlecit® Versus Oral Iron on Iron Deficient Chronic Kidney Disease (CKD) Patients Receiving Erythropoietic Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER0201
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-02

CONDITIONS: Anemia, Iron-Deficiency; Kidney Failure, Chronic
Keywords: Iron deficiency; Anemia; Chronic kidney disease; Erythropoietic agents; Sodium Ferric Gluconate; Anemia, Iron-Deficiency/drug therapy/etiology; Kidney Failure, Chronic/blood/complications/therapy; Erythropoietin, Recombinant/adverse effects/therapeutic use
MeSH Terms: conditions — Anemia, Iron-Deficiency; Kidney Failure, Chronic; Iron Deficiencies; Anemia; Renal Insufficiency, Chronic; Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — ferric gluconate; Sucrose; Iron-Dextran Complex

ARMS (2):
- IV iron (Experimental)
  Interventions: Drug: Sodium Ferric Gluconate complex in sucrose
- oral iron (Active Comparator)
  Interventions: Drug: Ferrous sulfate tablets

INTERVENTIONS:
Drug: Sodium Ferric Gluconate complex in sucrose — Sodium ferric gluconate complex in sucrose, 250 mg IV weekly for 4 doses
  Other Names: Ferrlecit
  Arms: IV iron
Drug: Ferrous sulfate tablets — ferrous sulfate 325 mg three times daily for 6 weeks
  Arms: oral iron

SUMMARY:
This study compares the effect of Ferrlecit® (a form of intravenous iron) to ferrous sulfate (a form of oral iron) in treating anemia and iron deficiency in chronic kidney disease patients who are receiving erythropoietic agents, such as Procrit® and Aranesp®.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe anemia
* Iron deficiency
* Moderate to severe chronic kidney disease
* Receiving therapy with erythropoietic agent

Exclusion Criteria:

* Receiving dialysis
* Known sensitivity to Ferrlecit® or any of its components
* Clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-04; Primary Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adel R Rizkala, PharmD, MS, Study Director — Watson Laboratories, Inc.
Locations (24):
- United States (23):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - Hines, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - St Louis, Missouri
  - Detroit, New York
  - Mineola, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Charlotte, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Fairfax, Virginia
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferrlecit: Sodium ferric gluconate complex in sucrose injection
Period: Overall Study
Arm/Group | Ferrlecit | Oral Iron
Started | 26 | 26
Completed | 20 | 20
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Did not meet lab incusion criteria | 2 | 3
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrlecit | Oral Iron | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 14 | 18 | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 67.4 (17.75) | 66.1 (14.65) | 66.8 (16.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Baseline Hemoglobin Concentration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferrlecit | Oral Iron
Number analyzed (Participants) | 24 | 24
g/dL | 10.3 (0.90) | 10.4 (0.92)

2. Secondary Outcome: Baseline Serum Ferritin Concentration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ferrlecit | Oral Iron
Number analyzed (Participants) | 24 | 24
ng/mL | 74.3 (80.95) | 68.7 (67.36)

3. Primary Outcome: Change in Hemoglobin (Hgb)
Description: Change from baseline to 7 weeks after 4 consecutive weekly Ferrlecit 250 mg intravenious infusion and change from baseline to 4 weeks after 6 weeks oral ferrous sulfate 325 mg tablets t.i.d.
Time Frame: Baseline to 10 weeks
Population: Modified ITT with LOCF imputation
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferrlecit | Oral Iron
Number analyzed (Participants) | 24 | 24
g/dL | 1.2 (1.23) | 1.0 (1.34)

4. Secondary Outcome: Change in Serum Ferritin
Description: as for outcome 3
Time Frame: Baseline to 10 weeks
Population: Modified ITT with LOCF imputation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ferrlecit | Oral Iron
Number analyzed (Participants) | 24 | 24
ng/mL | 150.0 (113.11) | 18.1 (33.66)

ADVERSE EVENTS:
Arm/Group | Ferrlecit | Oral Iron
Serious Adverse Events (participants affected / at risk) | 4/26 | 2/26
Other Adverse Events (participants affected / at risk) | 18/26 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrlecit (N=26) | Oral Iron (N=26)
Acerbation of Chronic Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain Chest (General disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Myocardiac Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Gout Attack (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrlecit (N=26) | Oral Iron (N=26)
Fever (General disorders) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 0 (0)
Accidental Injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Abdominal Pain (General disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Melena (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Edema (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Peripheral Edema (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Increase Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less